CLINICAL TRIAL: NCT00923845
Title: Low Intensity Allogeneic Hematopoietic Stem Cell Transplantation Therapy of Metastatic Renal Cell Carcinoma Using Early and Multiple Donor Lymphocyte Infusions Consisting of Sirolimus-Generated Donor Th2 Cells
Brief Title: Low-Intensity Stem Cell Transplantation With Multiple Lymphocyte Infusions to Treat Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Fowler, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080088; 08-C-0088; NCT00641485 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Renal Cell Carcinoma; Graft-Versus-Host Disease; Engraftment Syndrome
Keywords: Metastatic Renal Cell Carcinoma; Allogeneic Hematopoietic Stem Cell Transplant; Th2 Cells; Sirolimus; Pentostatin; Kidney Cancer; Renal Cell Carcinoma; Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Graft vs Host Disease; Kidney Neoplasms | interventions — Pentostatin; Sirolimus; Cyclophosphamide; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donors (Other): A sibling who is 6/6 HLA --matched with the recipient. Donors undergo donor lymphocyte harvest and stem cell mobilization and harvest.
  Interventions: Procedure: Donor Lymphocyte Harvest; Procedure: Donor Hematopoietic Stem Cell Harvest
- Recipients (Other): Recipients undergo induction therapy, allogeneic stem cell therapy and GVHD prophylaxis.
  Interventions: Drug: Pentostatin; Drug: Sirolimus; Drug: Cyclophosphamide; Procedure: Allogeneic Hematopoietic Stem Cell Transplant (HSCT); Procedure: Th2 rapa cells; Procedure: Induction Therapy; Procedure: GVHD prophylaxis

INTERVENTIONS:
Drug: Pentostatin — Pentostatin: 2- 4mg/m^2(CrCL based dosing) intravenous (IV) on days 1, 8, and 15
  Other Names: Nipent
  Arms: Recipients
Drug: Sirolimus — Sirolimus: 4 mg by mouth (PO) on days -3 to +7 post-transplant (No Sirolimus administered after day 7 post-stem cell transplant (SCT))
  Other Names: Rapamune
  Arms: Recipients
Drug: Cyclophosphamide — Cyclosporine: 2 mg/kg every 12 hours PO or IV starting on day -4 of hematopoietic stem cell transplant (HSCT)
  Other Names: Cytoxan
  Arms: Recipients
Procedure: Allogeneic Hematopoietic Stem Cell Transplant (HSCT) — Allogeneic Hematopoietic Stem Cell Transplant
  Arms: Recipients
Procedure: Th2 rapa cells — Th2 rapa cell Transplantation
  Arms: Recipients
Procedure: Donor Lymphocyte Harvest — Apheresis
  Arms: Donors
Procedure: Induction Therapy — Pentostatin and cyclophosphamide (PC) conditioning regimen.
  Arms: Recipients
Procedure: GVHD prophylaxis — Short course of sirolimus plus maintenance therapy with sirolimus A.
  Arms: Recipients
Procedure: Donor Hematopoietic Stem Cell Harvest — Following lymphocyte harvest, donors for recipients will undergo stem cell mobilization and harvest.
  Arms: Donors

SUMMARY:
Background:

Low-dose chemotherapy is easier for the body to tolerate than typical high-dose chemotherapy and involves a shorter period of complete immune suppression.

Donor immune cells called lymphocytes, or T cells, fight residual tumor cells that might have remained in the recipients body after stem cell transplant, in what is called a graft-versus-tumor (GVT) effect.

The immune-suppressing drug sirolimus appears to help prevent graft-versus-host disease (GVHD), a side effect of stem cell transplant in which donated T cells sometimes attack healthy tissues, damaging organs such as the liver, intestines and skin.

Th2 cells are cells collected from the transplant donor and grown in a high concentration of sirolimus.

Objectives:

To determine whether stem cell transplantation using low-dose chemotherapy and sirolimus-generated Th2 cells can cause a remission of advanced kidney cancer.

Eligibility:

Patients between 18 and 75 years of age who have kidney cancer that has spread beyond the kidney and who have a tissue-matched sibling stem cell donor.

Design:

Patients undergo stem cell transplantation as follows:

* Low-intensity chemotherapy with pentostatin and cyclophosphamide over a 21-day period to reduce the level of the immune system to prepare for the transplant. Pentostatin is given through a vein (intravenous (IV)) on days 1, 8 and 15; cyclophosphamide tablets are taken by mouth for 21 consecutive days.
* Sirolimus tablets, taken by mouth, starting 2 days before the transplant and continuing until 60 days after the transplant.
* IV infusions of stem cells and Th2 cells.

Following the transplant, patients have the following procedures:

* Additional Th2 cell infusions on days 14 and 45 after the transplant.
* Follow-up visits at the National Institutes of Health (NIH) Clinical Center twice a week for the first 6 months after the transplant and then less frequently for at least 5 years to evaluate response to treatment and treatment side effects. Evaluations include a bone marrow aspirate and biopsy 1 month after transplant and periodic blood tests and imaging procedures (e.g., computed tomography (CT) or magnetic resonance imaging (MRI) scans).

DETAILED DESCRIPTION:
Background:

Allogeneic hematopoietic stem cell transplantation (HSCT) represents a potentially effective treatment option for patients with metastatic renal cell carcinoma (RCC).

In a pilot clinical trial in refractory hematologic malignancy subjects, we have found that augmentation of a T cell-replete allograft with donor Th2 cells generated ex vivo in sirolimus (rapamycin; Th2.rapa cells) allows prompt donor engraftment after outpatient-intensity chemotherapy. This transplant approach has been associated with a low incidence of acute graft versus host disease (GVHD).

Based on these data, we seek to safely achieve objective clinical regression of metastatic RCC by the following new transplant approach. (1) The allograft will be administered after a low intensity, outpatient induction chemotherapy regimen consisting of pentostatin and cyclophosphamide. This regimen is intended to provide sufficient host immune T cell depletion, and as such, a conventional preparative regimen will not be administered. (2) To avoid mixed chimerism for rapid potentiation of graft-versus-tumor (GVT) effects, a growth colony stimulating factor (G-CSF) mobilized allograft will be augmented with donor lymphocyte infusion at day 14 post-transplant consisting of Th2.rapa cells.

Objectives:

Primary objective: (1) Determine whether this new, low-intensity transplant approach can yield objective partial or complete remission of metastatic RCC, with the goal of ruling out a partial response (PR)/complete response (CR) rate of 20% in favor of a rate of 60%.

Secondary objectives: (1) Evaluate the safety and immune-depleting properties of the pentostatin/cyclophosphamide regimen; (2) Characterize the engraftment kinetics and GVHD profile of this new transplant approach; and (3) Characterize post-transplant immunity in study subjects, including cytokine phenotype, immune reconstitution, and potential anti-tumor effector mechanisms.

Eligibility:

Adults (18 - 75 years) with metastatic RCC who have an eligible 6/6 human leukocyte antigen (HLA)-matched sibling donor.

Must have had one prior therapy with either sorafenib, sunitinib, or temsirolimus or any other Food and Drug Administration (FDA)-approved agent for therapy of metastatic renal cell carcinoma..

Life expectancy greater than or equal to 3 months, Karnofsky score greater than or equal to 80, relatively normal organ function, and absence of central nervous system (CNS) metastases.

Design:

Patients will receive a 21-day course of pentostatin (intravenous infusion on days 1, 8, and 15; 4 mg/m^2 per dose) and daily oral cyclophosphamide (200 mg per day).

Patients will receive a mobilized, T cell-replete allogeneic hematopoietic stem cell graft followed by a pre-emptive donor lymphocyte infusion with donor Th2 cells at day 14 post-transplant. GVHD prophylaxis will consist of a short-course of sirolimus plus maintenance therapy with cyclosporine A.

If greater than or equal to 2/5 partial or complete responses are observed within 6 months post-transplant, the therapy will be considered potentially promising, and will be expanded in a Simon two-stage design to evaluate a total of n = 14 subjects. If greater than or equal to 5/14 PR/CR are achieved, the therapy will be considered worthy of further investigation.

ELIGIBILITY:
* INCLUSION CRITERIA: Recipient

Diagnosis of metastatic renal cell carcinoma, either clear cell type or non-clear cell type. The diagnosis must be confirmed by the Laboratory of Pathology of National Cancer Institute (NCI) or Hackensack (there will be no central pathology review).

The consent process will include a discussion of the potential role of high-dose interleukin-2 (IL-2) therapy prior to protocol enrollment. High-dose IL-2 therapy is not widely available, but may be available on an NCI protocol (Dr. Yang) or through Dr. Alter for Hackensack patients. IL-2 therapy may also be administered by any other qualified physician; the Novartis web-site has a list of such physicians. For subjects who are deemed to be eligible for high-dose IL-2 and elect to receive this therapy, such subjects must have progressive disease post-IL-2 to enter this study; such subjects must also have received and have had progressive disease after therapy with one of the agents listed below.

Subject must have progressive disease after therapy consisting of one of the following Food and Drug Administration (FDA)-approved agents: sorafenib, sunitinib, or temsirolimus.

Patients 18 - 75 years of age. Subjects older than 75 will not be enrolled due to an increased rate of transplant-related complications.

Must have consenting sibling matched at 6/6 human leukocyte antigen (HLA) antigens (A, B, DR).

Patient or legal guardian must be able to give informed consent.

All previous therapy must be completed at least 2 weeks prior to study entry. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less.

Karnofsky performance status greater than or equal to 80%.

Life expectancy of at least 3 months.

Left ventricular ejection fraction greater than 40% (multi-gated acquisition scan (MUGA) or echo) within 28 days of enrollment.

Carbon monoxide diffusing capacity (DLCO) greater than 50% of expected value (hemoglobin (Hb) corrected), obtained within 28 days of enrollment.

Creatinine clearance greater than or equal to 40 ml/min. Creatinine clearance will be determined by testing of a 24 hour urine collection and simultaneous serum creatinine value. In previous studies, the creatine clearance of patients with metastatic renal cell cancer who underwent nephrectomy was 53 plus or minus 19.

Serum total bilirubin less than 2.5 mg/dl, and serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values less than or equal to 2.5 times the upper limit of normal. ALT and AST values above these levels may be accepted (up to a maximum of 5 times the upper limit of normal), at the discretion of the principal investigator (PI) or study chairperson, if such elevations are thought to be due to liver involvement by malignancy.

INCLUSION CRITERIA : Donor

Sibling who is 6/6 HLA-matched with recipient.

Ability to give informed consent.

Age 18 years to 80 years. Donors older than 80 will not be eligible due to potentially increased complications from the donation procedure.

Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.

Donors must be human immunodeficiency virus (HIV) negative, hepatitis B surface antigen negative, and hepatitis C antibody negative. This is to prevent the possible transmission of these infections to the recipient. Donors with a history of hepatitis B or hepatitis C infections may be eligible. However, eligibility determination of such patients will require a hepatology consultation. The risk/benefit of the transplant and the possibility of transmitting hepatitis will be discussed with the patient and eligibility will then be determined by the principal investigator.

A donor who is lactating must substitute formula feeding for her infant during the period of cytokine administration. Filgrastim may be secreted in human milk, although its bioavailability from this source is not known. Limited clinical data suggest that administration of filgrastim or to neonates is not associated with adverse outcomes.

EXCLUSION CRITERIA: Recipient

Active infection that is not responding to antimicrobial therapy.

Active central nervous system (CNS) involvement by malignancy.

HIV infection. There is theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.

Chronic active hepatitis B. Patient may be hepatitis B core antibody positive. For patients with concomitant positive hepatitis B surface antigen, patient will require a hepatology consultation. The risk/benefit profile of transplant and hepatitis B will be discussed with the patient and eligibility determined by the principal investigator and protocol chairperson.

Hepatitis C infection. Patient may have hepatitis C infection. However, each patient will require a hepatology consultation. The risk/benefit profile of transplant and hepatitis C will be discussed with the patient and eligibility determined by the principal investigator and protocol chairperson.

Pregnant or lactating. Patients of childbearing potential must use an effective method of contraception from the time of study entry to at least one year post-transplant; effective methods include intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation/hysterectomy, partner s vasectomy, or barrier methods (condom, diaphragm, or cervical cap). Males on the protocol, and their partners of child-bearing potential, must also use an effective form of contraception at study entry and for one year post-transplant. The effects of the chemotherapy, the subsequent transplant, and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to the infant; therefore, women should not breastfeed during the interval from study entry to one year post-transplant.

History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent (as determined by principal investigator or study chairman).

EXCLUSION CRITERIA: Donor

History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.

History of hypertension that is not controlled by medication, stroke, or severe heart disease. Individuals with symptomatic angina will be considered to have severe heart disease and will not be eligible to be a donor.

No other medical contraindications to stem cell donation (i.e. severe atherosclerosis, autoimmune disease, iritis or episcleritis, deep venous thrombosis, cerebrovascular accident). Patients with a history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis.

History of prior malignancy. However, cancer survivors who have undergone potentially curative therapy may be considered for stem cell donation on a case-by-case basis. The risk/benefit of the transplant and the possibility of transmitting viable tumor cells at the time of transplantation will be discussed with the patient.

Donors must not be pregnant. The effects of cytokine therapy on a fetus are unknown. Donors of childbearing potential must use an effective method of contraception from the time of study entry until at least one year post-transplant.

Anemia (Hb less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000 per microliter).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Fowler, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLaughlin JK, Lipworth L, Tarone RE. Epidemiologic aspects of renal cell carcinoma. Semin Oncol. 2006 Oct;33(5):527-33. doi: 10.1053/j.seminoncol.2006.06.010. PMID 17045081
- [Background] Shuch BM, Lam JS, Belldegrun AS, Figlin RA. Prognostic factors in renal cell carcinoma. Semin Oncol. 2006 Oct;33(5):563-75. doi: 10.1053/j.seminoncol.2006.06.006. PMID 17045085
- [Background] Patard JJ, Leray E, Rioux-Leclercq N, Cindolo L, Ficarra V, Zisman A, De La Taille A, Tostain J, Artibani W, Abbou CC, Lobel B, Guille F, Chopin DK, Mulders PF, Wood CG, Swanson DA, Figlin RA, Belldegrun AS, Pantuck AJ. Prognostic value of histologic subtypes in renal cell carcinoma: a multicenter experience. J Clin Oncol. 2005 Apr 20;23(12):2763-71. doi: 10.1200/JCO.2005.07.055. PMID 15837991
- [Result] Mossoba ME, Halverson DC, Kurlander R, Schuver BB, Carpenter A, Hansen B, Steinberg SM, Ali SA, Tageja N, Hakim FT, Gea-Banacloche J, Sportes C, Hardy NM, Hickstein DD, Pavletic SZ, Khuu H, Sabatini M, Stroncek D, Levine BL, June CH, Mariotti J, Rixe O, Fojo AT, Bishop MR, Gress RE, Fowler DH. High-Dose Sirolimus and Immune-Selective Pentostatin plus Cyclophosphamide Conditioning Yields Stable Mixed Chimerism and Insufficient Graft-versus-Tumor Responses. Clin Cancer Res. 2015 Oct 1;21(19):4312-20. doi: 10.1158/1078-0432.CCR-15-0340. Epub 2015 Jun 12. PMID 26071480
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0088.html

RESULTS

PARTICIPANT FLOW:
Period: Donor Lymphocyte Harvest
Arm/Group | Donors | Recipients
Started | 13 | 0
Completed | 13 | 0
Not Completed | 0 | 0
Period: Donor Hematopoietic Stem Cell Harvest
Arm/Group | Donors | Recipients
Started | 13 | 0
Completed | 13 | 0
Not Completed | 0 | 0
Period: Induction Therapy
Arm/Group | Donors | Recipients
Started | 0 | 12
Completed | 0 | 10
Not Completed | 0 | 2
Not completed — Poor performance status | 0 | 2
Period: Allogeneic Stem Cell Therapy
Arm/Group | Donors | Recipients
Started | 0 | 10
Received Each of 3 Planned T-Rapa DLI | 0 | 8
Received More Unmanipulated DLI for PD | 0 | 6
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donors | Recipients | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.14 (9.06) | 58.03 (8.01) | 55.48 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Clinical Regression of Metastatic Renal Cell Carcinoma (Partial Response (PR)) or Complete Remission of Tumor (Complete Response (CR))
Description: Response was assessed by computed tomography measurements and the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the largest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 Months Post-Transplant (Day +100)
Measure: Number; unit: participants
Groups:
- Recipient: Recipients undergo induction therapy, allogeneic stem cell therapy and GVHD prophylaxis.
Arm/Group | Recipient
Number analyzed (Participants) | 10
participants
  Partial Response (PR) | 0
  Complete Response (CR) | 0
  Progressive Disease (PD) | 8
  Stable Disease (SD) | 1
  Not Applicable (NA) | 1

2. Secondary Outcome: Count of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 50 months and 6 days
Measure: Count of Participants; unit: Participants
Groups:
- Donor: A sibling who is 6/6 HLA --matched with the recipient. Donors undergo donor lymphocyte harvest and stem cell mobilization and harvest.
Arm/Group | Donor | Recipient
Number analyzed (Participants) | 13 | 12
Participants | 0 | 12

3. Secondary Outcome: Count of Patients Having Neutropenia Attributable to the Pentostatin and Cyclophosphamide (PC) Regimen
Description: Absolute neutrophil count determination by complete blood count methodology (Absolute Neutrophil Count (ANC) < 500 Cells/µL).
Time Frame: During the 21-day PC regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Count of Patients Having an Infectious Complication Attributable to the Pentostatin and Cyclophosphamide (PC) Regimen
Description: Occurrence of infection by Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: During the 21-day PC regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Immune Depletion in Cluster of Differentiation 4 (CD4) Cells
Description: Reduction in cluster of differentiation 4 (CD4)+ T cells [change in median values and (range of values)].
Time Frame: Baseline and day 21 (completion of the pentostatin/cyclophosphamide regimen)
Measure: Median (Full Range); unit: Cells/µL
Arm/Group | Recipient
Number analyzed (Participants) | 10
Cells/µL
  Baseline | 503 [124 to 1487]
  Day 21 | 54 [10 to 107]

6. Secondary Outcome: Immune Depletion in Cluster of Differentiation 8 (CD8)+ T Cells
Description: Reduction in cluster of differentiation 8 (CD8)+ T cells [change in median values and (range of values)].
Time Frame: Baseline and day 21 (completion of the pentostatin/cyclophosphamide regimen)
Measure: Median (Full Range); unit: cells/µL
Arm/Group | Recipient
Number analyzed (Participants) | 10
cells/µL
  Baseline | 239 [56 to 770]
  Day 21 | 45 [12 to 131]

7. Secondary Outcome: Immune Suppression
Description: Immune suppression is defined by the frequency of elimination of a pre-transplant T cell cytokine value.
Time Frame: Cytokine analysis at baseline and within 24 hours of completion of the pentostatin/cyclophosphamide regimen
Measure: Number; unit: % of undetectable cytokine measurements
Arm/Group | Recipient
Number analyzed (Participants) | 10
% of undetectable cytokine measurements
  Positive at baseline | 100
  Negative at baseline | 0
  Positive 24 hours after regimen | 0
  Negative 24 hours after regimen | 100

8. Secondary Outcome: Engraftment Donor T Cell and Myeloid Cell Chimerism
Description: Donor Genetic Elements by variable number tandem repeat-polymerase chain reaction (VNTR-PCR) Analysis.
Time Frame: Days 14, 28, 45, and 60 post transplant
Measure: Median (Full Range); unit: Percent Donor by VNTR-PCR Analysis
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percent Donor by VNTR-PCR Analysis
  Day 14 donor T cell chimerism | 61 [7 to 77]
  Day 28 donor T cell chimerism | 72 [9 to 91]
  Day 45 donor T cell chimerism | 74 [21 to 88]
  Day 60 donor T cell chimerism | 77 [26 to 95]
  Day 14 myeloid cell chimerism | 0 [0 to 27]
  Day 28 myeloid cell chimerism | 13 [4 to 50]
  Day 45 myeloid cell chimerism | 18 [11 to 67]
  Day 60 myeloid cell chimerism | 26 [13 to 76]

9. Secondary Outcome: Count of Patients With Grade II or Greater Acute Graft Versus Host Disease (GVHD) in First 100 Days Post-Transplant
Description: Acute GVHD is assessed by the 1994 Consensus Conference on Acute GVHD grading criteria. Acute GVHD may include rash, diarrhea, and liver damage (i.e. rash Grading: <25% body surface area (BSA) = 1, rash 25-50% BSA = 2, generalized erythroderma = 3, and desquamation and bullae = 4); liver Grading: total bilirubin 2-3 mg/dl = 1, total bilirubin 3-6 mg/dl =2, total bilirubin 6-15 mg/dl =3, and total bilirubin >15 mg/dl = 4)).
Time Frame: 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 12
Participants | 0

10. Secondary Outcome: Count of Patients With Late Acute Graft Versus Host Disease (GVHD) After Day 100 Post-Transplant
Description: Acute GVHD is assessed by the 1994 Consensus Conference on Acute GVHD grading criteria. Acute GVHD is assessed by the 1994 Consensus Conference on Acute GVHD grading criteria. Acute GVHD may include rash, diarrhea, and liver damage (i.e. rash Grading: <25% body surface area (BSA) = 1, rash 25-50% BSA = 2, generalized erythroderma = 3, and desquamation and bullae = 4); liver Grading: total bilirubin 2-3 mg/dl = 1, total bilirubin 3-6 mg/dl =2, total bilirubin 6-15 mg/dl =3, and total bilirubin >15 mg/dl = 4)).
Time Frame: 100 days post-transplant through 5 years post-transplant
Population: Only 6 patients were evaluable for this endpoint due to death due to malignancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 6
Participants | 4

11. Secondary Outcome: Count of Patients With Chronic Graft Versus Host Disease (GVHD)
Description: Chronic GVHD was assessed by the 2005 Chronic GVHD Consensus Project. Chronic GVHS may include dryness of the mouth and eyes, weight loss, liver damage and lung damage leading to cough and shortness of breath (i.e. skin Grading: no symptoms = 0, <18% body surface area (BSA) = 1, 19-50% BSA = 2, and >50% BSA = 3); oral cavity Grading: no symptoms = 0, mild symptoms = 1, moderate symptoms =2 and severe symptoms =3)).
Time Frame: For the duration of post-transplant follow-up
Population: Only 4 patients were evaluable due to mortality from malignancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient
Number analyzed (Participants) | 4
Participants | 1

12. Secondary Outcome: Cluster of Differentiation 4 (CD4) T Cells Immune Reconstitution
Description: CD4 T Cells immune reconstitution is defined as distribution of CD4+ T cells subsets within naïve, central memory, effector memory, and effector memory-RA cells analyzed by flow cytometry.
Time Frame: Days 14, 60, and 100 post transplant
Population: The values for each subset were stable at days 60 and 100 relative to day 14 values.
Measure: Median (Standard Deviation); unit: Percentage of total CD4 cell subsets
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percentage of total CD4 cell subsets
  Day 14 | 22 (3)
  Day 60 | 20 (2)
  Day 100 | 19 (2)

13. Secondary Outcome: Cluster of Differentiation 8 (CD8)+ T Cells Immune Reconstitution
Description: CD8+ T Cells immune reconstitution is defined as distribution of CD8+ T cells subsets within naïve, central memory, effector memory, and effector memory-RA cells analyzed by flow cytometry.
Time Frame: Days 14, 60, and 100 post transplant
Population: The values for each subset were stable at days 60 and 100 relative to day 14 values.
Measure: Median (Standard Deviation); unit: Percent of total CD8 cell subsets
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percent of total CD8 cell subsets
  Day 14 | 6 (1)
  Day 60 | 5 (1)
  Day 100 | 4 (1)

14. Secondary Outcome: Percentage of Cluster of Differentiation 4 (CD4)+ T Cells Expressing the Th2 Transcription Factor GATA Binding Protein 3 (GATA-3)
Description: Intra-cellular flow cytometry detection of GATA3 transcription factor.
Time Frame: Days 14, 60 and 100 post transplant
Population: The values for each subset were stable at days 60 and 100 relative to day 14 values.
Measure: Median (Full Range); unit: Percentage of total CD4+ T cells
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percentage of total CD4+ T cells
  Day 14 | 42 [31 to 64]
  Day 60 | 37 [28 to 44]
  Day 100 | 43 [20 to 49]

15. Secondary Outcome: Percentage of Cluster of Differentiation 4 (CD4)+ T Cells Expressing the Th1 Transcription Factor T-bet
Description: CD4+ T cells were analyzed by flow cytometry for intracellular detection of Tbet transcription factor.
Time Frame: Days 14, 60, and 100 post transplant
Population: The values for each subset were stable at days 60 and 100 relative to day 14 values.
Measure: Median (Full Range); unit: Percentage of total CD4+T cells
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percentage of total CD4+T cells
  Day 14 | 8 [3 to 16]
  Day 60 | 8 [1 to 17]
  Day 100 | 6 [2 to 19]

16. Secondary Outcome: Percentage of Cluster of Differentiation 4 (CD4)+ T Cells Expressing the T-reg Transcription Factor Forkhead Box P3 (FoxP3))
Description: CD4+ T cells were analyzed by flow cytometry for intracellular expression of FoxP3.
Time Frame: Days 14, 60, and 100 post transplant
Population: The values for each subset were stable at days 60 and 100 relative to day 14 values.
Measure: Median (Full Range); unit: Percentage of total CD4+ T cells
Arm/Group | Recipient
Number analyzed (Participants) | 10
Percentage of total CD4+ T cells
  Day 14 | 8 [4 to 14]
  Day 60 | 6 [1 to 13]
  Day 100 | 3 [1 to 10]

ADVERSE EVENTS:
Time Frame: 50 months and 6 days
Arm/Group | Donor | Recipient
All-Cause Mortality (participants affected / at risk) | 0/13 | 7/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 8/12
Other Adverse Events (participants affected / at risk) | 0/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor (N=13) | Recipient (N=12)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 0 (0) | 2 (2)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 0 (0) | 5 (5)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor (N=13) | Recipient (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 0 (0) | 5 (18)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 0 (0) | 6 (44)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Adrenal insufficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Hepatobiliary disorders) | 0 (0) | 5 (15)
Alkaline phosphatase (Hepatobiliary disorders) | 0 (0) | 2 (3)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Amylase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac General - Other (Cardiac disorders) | 0 (0) | 2 (4)
Confusion (Nervous system disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Edema: limb (Cardiac disorders) | 0 (0) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 5 (5)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 2 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Growth and Development - Other (General disorders) | 0 (0) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 9 (61)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Hemorrhage, GI::Cecum/appendix (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Liver (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 0 (0) | 2 (3)
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection - Other (Infections and infestations) | 0 (0) | 2 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Ungual (nails) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Renal and urinary disorders) | 0 (0) | 2 (3)
Infection with unknown ANC::Blood (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection with unknown ANC::Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection with unknown ANC::Trachea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 8 (43)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Mood alteration::Depression (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Neurology - Other (Nervous system disorders) | 0 (0) | 4 (4)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 6 (25)
Ocular/Visual - Other (Eye disorders) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Pain - Other (General disorders) | 0 (0) | 5 (5)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain::Buttock (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Pain NOS (General disorders) | 0 (0) | 2 (2)
Pain::Pelvis (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 8 (25)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 5 (60)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 (0) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 7 (34)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Cardiac disorders) | 0 (0) | 1 (1)
Syndromes - Other (General disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Cardiac disorders) | 0 (0) | 4 (5)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (12)
Weight loss (General disorders) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No